CLINICAL TRIAL: NCT05100069
Title: General Use-results Survey of Alunbrig Tablets "Non-small Cell Lung Cancer"
Brief Title: Survey of Brigatinib Used To Treat People With Non-Small Cell Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: C25026; jRCT2031210404 (Registry Identifier: jRCT)
Record Dates: First submitted 2021-10-28; First posted 2021-10-29 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — brigatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Brigatinib Tablets: Brigatinib 90 milligrams (mg), tablet, orally, once daily for up to 7 days, followed by 180 mg, tablets, once daily for 51 weeks. Participants received interventions as part of routine medical care.
  Interventions: Drug: Brigatinib

INTERVENTIONS:
Drug: Brigatinib — Brigatinib Tablets
  Other Names: Alunbrig Tablets

SUMMARY:
This study is a survey in Japan of Brigatinib tablets used to treat Japanese people with non-small cell lung cancer. The study sponsor will not be involved in how the participants are treated but will provide instructions on how the clinics will record what happens during the study.

The main aim of the study is to check for side effects related to lung disease from Brigatinib. During the study, participants with non-small cell lung cancer will take Brigatinib tablets according to their clinic's standard practice. The study doctors will check for side effects from Brigatinib for 1 year.

ELIGIBILITY:
Inclusion criteria Participants with unresectable advanced/recurrent ALK fusion gene-positive non-small cell lung cancer.

Exclusion criteria Participants who has a history of hypersensitivity to any component of birigatinib.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with unresectable advanced/recurrent ALK fusion gene-positive non-small cell lung cancer.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events Related to Interstitial Lung Disease | Up to 1 year
  An adverse event (AE) is any untoward or undesirable medical occurrence in a participant linked in time with the use of a pharmaceutical/ medicinal product. They are not limited to the events with clear causal relationship with treatment with concerned drug. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda Selected Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/6182c950eb0e19002afd69fa